CLINICAL TRIAL: NCT04156620
Title: A Randomized, Double-blind, Placebo-controlled, Parallel Group, Phase III Multicenter Study of Intravenous Secukinumab to Compare Efficacy at 16 Weeks With Placebo and to Assess Safety and Tolerability up to 52 Weeks in Subjects With Active Ankylosing Spondylitis or Non-radiographic Axial SpondyloArthritis
Brief Title: Study to Demonstrate the Efficacy, Safety and Tolerability of an Intravenous Regimen of Secukinumab Compared to Placebo in Subjects With Active axSpA
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: CAIN457P12301
Record Dates: First submitted 2019-10-08; First posted 2019-11-07 (Actual); Results first posted 2024-01-23 (Actual); Last update posted 2024-06-18 (Actual); Status verified 2024-06

CONDITIONS: Ankylosing Spondylitis
Keywords: Active axSpA; Axial spondyloarthritis; non-radiographic-axSpA; nr-axSpA; ankylosing spondylitis; AS; inflammatory back pain; sacroiliitis
MeSH Terms: conditions — Spondylitis, Ankylosing; Axial Spondyloarthritis; Non-Radiographic Axial Spondyloarthritis; Sacroiliitis | interventions — secukinumab

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: This is a double-blind, randomized treatment trial. Subjects, investigators, investigator staff and persons performing the assessments, will remain blind to the identity of the treatment from the time of randomization until database lock, using the following methods: (1) Randomization data are kept strictly confidential until the time of unblinding and will not be accessible by anyone else involved in the study with the exception of the bioanalyst, (2) the identity of the treatments will be concealed by the use of study treatment in form of vials, filled with secukinumab or placebo that are identical in appearance.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Secukinumab (Experimental): Secukinumab intravenous (i.v.) regimen
  Interventions: Drug: Secukinumab
- Placebo (Placebo Comparator): Placebo intravenous (i.v.) regimen
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Secukinumab — The subjects will receive secukinumab 6 mg/kg i.v. at randomization (Baseline (BSL) visit), followed by the administration of secukinumab 3 mg/kg i.v. every four weeks starting at Week 4 through Week 48 (exposure through Week 52)
  Other Names: AIN457
  Arms: Secukinumab
Drug: Placebo — The subjects will receive i.v. placebo at randomization (BSL visit), Weeks 4, 8, and 12 , followed by the administration of secukinumab 3 mg/kg i.v. at Week 16 and every four weeks through Week 48 (exposure through Week 52)
  Arms: Placebo

SUMMARY:
The purpose of this global study was to demonstrate the efficacy, safety, and tolerability of an intravenous (i.v.) regimen of secukinumab compared to placebo in participants with active ankylosing spondylitis (AS) or non-radiographic axial spondyloarthritis (nr-axSpA ) at Week 16 despite current or previous non-steroidal anti inflammatory drugs (NSAID), disease-modifying antirheumatic drugs (DMARD) and/or anti Tumor Necrosis Factor (TNF) therapy. In addition, to further support efficacy and safety of an i.v. regimen, data was collected for up to 52 weeks of treatment.

DETAILED DESCRIPTION:
This multicenter study used a randomized, double-blind, placebo-controlled, parallel-group design to study the efficacy, safety, and tolerability of treatment with intravenous secukinumab (initial dose of 6 mg/kg followed thereafter with 3 mg/kg administered every four weeks starting at Week 4) in subjects with active axial spondyloarthritis (axSpA). The study population consisted of active of 413 participants with AS and 113 participants with active nr-axSpA.

This study consisted of 4 periods totaling up to 70 weeks: the screening period (up to 10 weeks), the treatment period 1 (total duration of 16 weeks), treatment period 2 (total duration of 36 weeks) followed by the safety follow up period of 8 weeks after the end of treatment visit (at Week 60) regardless of whether participant completed the study as planned or discontinued prematurely.

At baseline, participants were randomized to one of the two treatment groups and stratified to disease condition (AS or nr-axSPa):

* Group 1: secukinumab 6 mg/kg i.v.) at baseline and which was followed by the administration of secukinumab 3 mg/kg i.v. every four weeks starting at Week 4 through Week 48 (exposure through Week 52) at clinic visits
* Group 2: i.v. placebo at baseline, Weeks 4, 8, and 12 and switched to secukinumab 3 mg/kg i.v. at Week 16 and every four weeks through Week 48 (exposure through Week 52) at clinic visits

Although study treatment was open label secukinumab i.v. starting at Week 16, all subjects and investigators/site staff remained blinded to original treatment assignment to ensure unbiased efficacy and safety assessments for the remainder of the study. This study enrolled participants with active disease despite current or previous NSAIDs, conventional DMARDs and/or TNF inhibitor therapy or intolerance to these therapies. The regular assessment of disease activity ensured that subjects who experienced worsening of disease in any of the treatment groups could exit the study at any time upon their own accord or based on the advice of the investigator.

A temporary pause of study recruitment only was implemented from 09-Apr-2020 to 11-May-2020, due to the COVID-19 pandemic, but not for study visits, assessments or other conduct of the study.

ELIGIBILITY:
Inclusion Criteria:

Subjects eligible for inclusion in this study must meet all of the following criteria:

1. Subject must be able to understand and communicate with the investigator, comply with the requirements of the study. and must give written, signed and dated informed consent before any study assessment is performed
2. Male and non-pregnant, non-lactating female patients ≥ 18 years of age
3. Diagnosis of axSpA according to ASAS criteria

   1. Inflammatory back pain for at least 6 months
   2. Onset before 45 years of age
4. For subjects with AS: Diagnosis of AS with prior documented radiologic evidence (x-ray or radiologist's report) fulfilling the Modified New York criteria for AS
5. For subjects with nr-axSpA:

   X-ray of SIJ negative (centrally read) for AS by Modified NY criteria AND
   1. Sacroiliitis on MRI (centrally read) with ≥ 1 SpA feature OR HLA-B-27 positive with ≥2 SpA features AND
   2. Objective signs of inflammation at screening, evident by either MRI with SIJ inflammation (centrally read) AND / OR hsCRP > ULN (as defined by the central lab)
6. Active axial SpA assessed by BASDAI ≥4 cm (0-10 cm) at Baseline
7. Spinal pain as measured by BASDAI question #2 ≥ 4 cm (0-10 cm) at Baseline
8. Total back pain as measured by VAS ≥ 40 mm (0-100 mm) at Baseline
9. Subjects should have had inadequate response or failure to respond to at least 2 NSAIDs at an approved dose for a minimum of 4 weeks in total and a minimum of 2 weeks for each NSAID prior to randomization, or less than 4 weeks if therapy had to be withdrawn due to intolerance, toxicity or contraindications
10. Subjects who are regularly taking NSAIDs (including COX-1 or COX-2 inhibitors) as part of their AS or nr-axSpA therapy are required to be on a stable dose for at least 2 weeks before randomization
11. Subjects who are intolerant or have been inadequate responders to a TNF inhibitor (not more than one) will be allowed to enter into the study (not more than 20% per group). They must have experienced an inadequate response to previous or current treatment at an approved dose for at least 3 months prior to randomization, or have been intolerant to at least one administration of an anti-TNF agent. These subjects will undergo an appropriate wash-out period prior to randomization, if required

    1. 4 weeks for Enbrel® (etanercept) - with a terminal half-life of 102 ± 30 hours
    2. 8 weeks for Remicade® (infliximab) - with a terminal half-life of 8.0-9.5 days
    3. 10 weeks for Humira® (adalimumab) - with a terminal half-life of 10-20 days (average 2 weeks)
    4. 10 weeks for Simponi® (golimumab) - with a terminal half-life of 11-14 days
    5. 10 weeks for Cimzia® (certolizumab) - with a terminal half-life of 14 days
12. Subjects taking methotrexate (MTX) (≤ 25 mg/week ) or sulfasalazine (≤ 3 g/day) are allowed to continue their medication and must have taken it for at least 3 months and have to be on a stable dose for at least 4 weeks prior to randomization. Subjects on MTX must be on folic acid supplementation before randomization
13. Subjects who are on a conventional DMARD other than MTX or sulfasalazine must discontinue the DMARD 4 weeks prior to randomization, except for leflunomide, which must be be discontinued 8 weeks prior to randomization, unless a cholestyramine washout has been performed
14. Subjects taking systemic corticosteroids must be on a stable dose of ≤10 mg/day prednisone or equivalent for at least 2 weeks before randomization

Exclusion Criteria:

Subjects meeting any of the following criteria are not eligible for inclusion in this study

1. Subjects with total ankylosis of the spine
2. Chest x-ray or MRI with evidence of ongoing infectious or malignant process obtained within 3 months of screening and evaluated by a qualified physician
3. Subjects taking moderate and high potency opioid analgesics (e.g. methadone, hydromorphone, morphine)
4. Presence of significant medical problems which at investigator's discretion, will prevent the subject from participating in the study, including but not limited to the following: Subjects with severely reduced kidney function (estimated glomerular filtration rate (eGFR) <29 ml/min/1.73m2), history of renal trauma, glomerulonephritis, or patients with one kidney only, or a serum creatinine level exceeding 1.5 mg/dl (132.6 μmol/L)
5. Any therapy by intra-articular injections (e.g. corticosteroid) within 4 weeks before Randomization
6. Underlying conditions (including, but not limited to metabolic, hematologic, renal, hepatic, pulmonary, neurologic, endocrine, cardiac, infectious or gastrointestinal) which in the opinion of the investigator significantly immunocompromises the subject and/or places the subject at unacceptable risk for receiving an immunomodulatory therapy
7. Any medical or psychiatric condition which, in the Investigator's opinion, would preclude the participant from adhering to the protocol or completing the study per protocol
8. Active systemic infections during the last two weeks (exception: common cold) prior to randomization or any infection that reoccurs on a regular basis
9. History of ongoing, chronic or recurrent infectious disease or evidence of tuberculosis infection as defined by either a positive purified protein derivative (PPD) skin test (the size of induration will be measured after 48-72 hours, and a positive result is defined as an induration of ≥ 5 mm or according to local practice/guidelines) or a positive QuantiFERON TB-Gold test as indicated in the assessment schedule in Table 8-1. Subjects with a positive test may participate in the study if further work up (according to local practice/guidelines) establishes conclusively that the subject has no evidence of active tuberculosis. If presence of latent tuberculosis is established, then treatment according to local country guidelines must have been initiated
10. Past medical history of infection with HIV or hepatitis B prior to randomization or active infection or on treatment for Hepatitis C at randomization
11. History of lymphoproliferative disease or any known malignancy, or history of malignancy of any organ system treated or untreated within the past 5 years, regardless of whether there is evidence of local recurrence or metastases (except for skin Bowen's disease, or basal cell carcinoma or actinic keratoses that have been treated with no evidence of recurrence in the past 12 weeks; carcinoma in situ of the cervix or non-invasive malignant colon polyps that have been removed)
12. Use or planned use of prohibited concomitant medication (see Section 6.2.2)
13. Inability or unwillingness to undergo repeated venipuncture (e.g., because of poor tolerability or lack of access to veins)
14. Pregnant or nursing (lactating) women, where pregnancy is defined as the state of a female after conception and until the termination of gestation, confirmed by a positive hCG laboratory test
15. History or evidence of ongoing alcohol or drug abuse, within the last six months before randomization
16. Screening total WBC count <3,000/μl, or platelets <100,000/μl or neutrophils <1,500/μl or hemoglobin <8.5 g/dl (85 g/L)
17. History of clinically significant liver disease or liver injury indicated by abnormal liver function tests, such as SGOT (AST), SGPT (ALT), alkaline phosphatase and serum bilirubin. The investigator should be guided by the following criteria:

    * Any single parameter may not exceed 2 x the upper limit of normal (ULN). A single parameter elevated up to and including 2 x ULN should be re-checked once more as soon as possible, and in all cases, at least prior to randomization, to rule-out laboratory error.
    * If the total bilirubin concentration is increased above 2 x ULN, total bilirubin should be differentiated into the direct and indirect reacting bilirubin. In any case, serum bilirubin should not exceed the value of 1.6 mg/dL (27 µmol/L)
18. Significant medical problems or diseases, including but not limited to the following:

    uncontrolled hypertension (≥160/95 mmHg), congestive heart failure (New York Heart Association status of class III or IV), uncontrolled diabetes, or very poor functional status precluding ability to perform self-care
19. Plans for administration of live vaccines during the study period or within 6 weeks prior to randomization
20. Women of child-bearing potential, defined as all women physiologically capable of becoming pregnant, unless they are using effective methods of contraception during the entire study or longer if required by locally approved prescribing information (e.g., 20 weeks in EU). Effective contraception methods include:

    * Total abstinence (when this is in line with the preferred and usual lifestyle of the subject. Periodic abstinence (e.g., calendar, ovulation, symptothermal, post-ovulation methods) and withdrawal are not acceptable methods of contraception
    * Female sterilization (have had surgical bilateral oophorectomy with or without hysterectomy) or tubal ligation at least six weeks before taking study treatment. In case of oophorectomy alone, only when the reproductive status of the woman has been confirmed by follow up hormone level assessment
    * Male sterilization (at least 6 months prior to screening). For female subjects on the study, the vasectomized male partner should be the sole partner for that subject
    * Barrier methods of contraception: Condom or Occlusive cap (diaphragm or cervical/vault caps). For UK: with spermicidal foam/gel/film/cream/ vaginal suppository
    * Use of oral, injected or implanted hormonal methods of contraception or other forms of hormonal contraception that have comparable efficacy (failure rate <1%), for example hormone vaginal ring or transdermal hormone contraception
    * Placement of an intrauterine device or intrauterine system In case of use of oral contraception women should have been stable on the same pill for a minimum of 3 months before taking study treatment.

    Women are considered post-menopausal and not of child bearing potential if they have had 12 months of natural (spontaneous) amenorrhea with an appropriate clinical profile (e.g., age appropriate, history of vasomotor symptoms) or have had surgical bilateral oophorectomy (with or without hysterectomy) or tubal ligation at least six weeks prior to randomization. In the case of oophorectomy alone, only when the reproductive status of the woman has been confirmed by follow up hormone level assessment is she considered not of childbearing potential.
21. Active ongoing inflammatory diseases other than axSpA that might confound the evaluation of the benefits of secukinumab therapy, including inflammatory bowel disease or uveitis
22. Current severe progressive or uncontrolled disease which in the judgment of the clinical investigator renders the subject unsuitable for the trial
23. Use of other investigational drugs at the time of enrollment, or within 5 half- lives of enrollment, or within 4 weeks until the expected pharmacodynamic effect has returned to baseline, whichever is longer; or longer if required by local regulations
24. History of hypersensitivity to any of the study drug constituents
25. Previous exposure to secukinumab (AIN457) or any other biologic drug directly targeting IL-17 or the IL-17 receptor
26. Previous treatment with any cell-depleting therapies including but not limited to anti-CD20 or investigational agents (e.g., CAMPATH, anti-CD4, anti-CD5, anti-CD3, anti-CD19)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 527 (Actual)
Dates: Start 2019-12-11 (Actual); Primary Completion 2022-02-17 (Actual); Study Completion 2022-12-20 (Actual)

CONTACTS AND LOCATIONS:
Locations (91):
- United States (25):
  - Novartis Investigative Site, Irvine, California
  - Novartis Investigative Site, La Mesa, California
  - Novartis Investigative Site, San Leandro, California
  - Novartis Investigative Site, Upland, California
  - Novartis Investigative Site, Ocoee, Florida
  - Novartis Investigative Site, Plantation, Florida
  - Novartis Investigative Site, Winter Park, Florida
  - Novartis Investigative Site, Bowling Green, Kentucky
  - Novartis Investigative Site, Cumberland, Maryland
  - Novartis Investigative Site, Grand Blanc, Michigan
  - Novartis Investigative Site, Lincoln, Nebraska
  - Novartis Investigative Site, Potsdam, New York
  - Novartis Investigative Site, Greensboro, North Carolina
  - Novartis Investigative Site, Middleburg Heights, Ohio
  - Novartis Investigative Site, Portland, Oregon
  - Novartis Investigative Site, Duncansville, Pennsylvania
  - Novartis Investigative Site, Columbia, South Carolina
  - Novartis Investigative Site, Jackson, Tennessee
  - Novartis Investigative Site, Memphis, Tennessee
  - Novartis Investigative Site, Katy, Texas
  - Novartis Investigative Site, Spring, Texas
  - Novartis Investigative Site, The Woodlands, Texas
  - Novartis Investigative Site, Everett, Washington
  - Novartis Investigative Site, Spokane, Washington
  - Novartis Investigative Site, Beckley, West Virginia
- Belgium (2):
  - Novartis Investigative Site, Brussels
  - Novartis Investigative Site, Leuven
- Brazil (6):
  - Novartis Investigative Site, Vitória, Espírito Santo
  - Novartis Investigative Site, Salvador, Estado de Bahia
  - Novartis Investigative Site, Juiz de Fora, Minas Gerais
  - Novartis Investigative Site, São Paulo, São Paulo
  - Novartis Investigative Site, Rio de Janeiro
  - Novartis Investigative Site, São José do Rio Preto
- Bulgaria (3):
  - Novartis Investigative Site, Pleven
  - Novartis Investigative Site, Plovdiv
  - Novartis Investigative Site, Sofia
- Colombia (6):
  - Novartis Investigative Site, Barranquilla, Atlántico
  - Novartis Investigative Site, Bucaramanga, Santander Department
  - Novartis Investigative Site, Ibagué, Tolima Department
  - Novartis Investigative Site, Barranquilla
  - Novartis Investigative Site, Bogotá
  - Novartis Investigative Site, Cundinamarca
- Czechia (3):
  - Novartis Investigative Site, Ostrava, Czech Republic
  - Novartis Investigative Site, Prague
  - Novartis Investigative Site, Uherské Hradiště
- Greece (2):
  - Novartis Investigative Site, Athens
  - Novartis Investigative Site, Pátrai
- Novartis Investigative Site, Guatemala City, Guatemala
- India (6):
  - Novartis Investigative Site, Surat, Gujarat
  - Novartis Investigative Site, Bangalore, Karnataka
  - Novartis Investigative Site, Mumbai, Maharashtra
  - Novartis Investigative Site, Nashik, Maharashtra
  - Novartis Investigative Site, Hyderabad, Telangana
  - Novartis Investigative Site, New Delhi
- Italy (2):
  - Novartis Investigative Site, Siena, SI
  - Novartis Investigative Site, Verona, VR
- Malaysia (5):
  - Novartis Investigative Site, Seremban, Negeri Sembilan
  - Novartis Investigative Site, Ipoh, Perak
  - Novartis Investigative Site, Kuching, Sarawak
  - Novartis Investigative Site, Kuala Lumpur
  - Novartis Investigative Site, Selangor Darul Ehsan
- Philippines (4):
  - Novartis Investigative Site, Lipa City, Batangas
  - Novartis Investigative Site, Dasmariñas, Cavite
  - Novartis Investigative Site, Manila
  - Novartis Investigative Site, Quezon
- Poland (5):
  - Novartis Investigative Site, Bialystok
  - Novartis Investigative Site, Krakow
  - Novartis Investigative Site, Sochaczew
  - Novartis Investigative Site, Torun
  - Novartis Investigative Site, Warsaw
- Russia (10):
  - Novartis Investigative Site, Chelyabinsk
  - Novartis Investigative Site, Kazan'
  - Novartis Investigative Site, Kemerovo
  - Novartis Investigative Site, Moscow
  - Novartis Investigative Site, Novosibirsk
  - Novartis Investigative Site, Petrozavodsk
  - Novartis Investigative Site, Saint Petersburg
  - Novartis Investigative Site, Ulyanovsk
  - Novartis Investigative Site, Yaroslavl
  - Novartis Investigative Site, Yekaterinburg
- South Korea (2):
  - Novartis Investigative Site, Gwangju
  - Novartis Investigative Site, Seoul
- Sweden (2):
  - Novartis Investigative Site, Danderyd
  - Novartis Investigative Site, Stockholm
- Thailand (4):
  - Novartis Investigative Site, Bangkoknoi, Bangkok
  - Novartis Investigative Site, Songkhla, Hat Yai
  - Novartis Investigative Site, Khon Kaen, THA
  - Novartis Investigative Site, Bangkok
- Turkey (Türkiye) (3):
  - Novartis Investigative Site, Adana
  - Novartis Investigative Site, Ankara
  - Novartis Investigative Site, Istanbul

IPD SHARING:
Plan to Share IPD: Yes
Novartis is committed to sharing access to patient-level data and supporting clinical documents from eligible studies with qualified external researchers. Requests are reviewed and approved by an independent review panel on the basis of scientific merit. All data provided is anonymized to protect the privacy of patients who have participated in the trial in line with applicable laws and regulations.
  This trial data availability is according to the criteria and process described on www.clinicalstudydatarequest.com
URL: https://clinicalstudydatarequest.com/Default.aspx

REFERENCES:
- See also: Patient Lay Trial Summary — https://www.novctrd.com/ctrdweb/patientsummary/patientsummaries?patientSummaryId=1809

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: 769 participants were screened for the study and 527 participants were randomized. However, one participant was mis-randomized and discontinued prior to dosing and is not included in the table below.
Groups:
- AIN457 6 mg/kg - 3 mg/kg i.v.: Participants received AIN457 (secukinumab) 6 mg/kg i.v. at baseline, followed by AIN457 3 mg/kg i.v. every four weeks starting at Week 4 through Week 48 (exposure through Week 52)
- Placebo - AIN457 3 mg/kg i.v.: Participants received i.v. placebo at baseline visit, Weeks 4, 8, and 12, followed by AIN457 (secukinumab) 3 mg/kg i.v. at Week 16 and every four weeks through Week 48 (exposure through Week 52)
Period: Overall Study
Arm/Group | AIN457 6 mg/kg - 3 mg/kg i.v. | Placebo - AIN457 3 mg/kg i.v.
Started | 264 | 262
Completed Period 1 (Baseline up to Week 16) | 255 | 253
Started Period 2 (Week 16 up Week 52) | 255 | 251 (2 patients completed Period 1 but discontinued prior to Period 2)
Completed Period 2 | 233 | 235
Completed (Completed up to Week 60 (follow-up)) | 227 | 233
Not Completed | 37 | 29
Not completed — Adverse event - TP 1 | 5 | 2
Not completed — Lost to follow-up TP 1 | 1 | 1
Not completed — Progressive disease - TP 1 | 0 | 1
Not completed — Subject decision - TP 1 | 3 | 5
Not completed — Adverse event - TP 2 | 5 | 6
Not completed — Death - TP 2 | 1 | 0
Not completed — Lost to follow-up - TP 2 | 5 | 2
Not completed — Physician decision - TP 2 | 4 | 2
Not completed — Pregnancy - TP 2 | 1 | 1
Not completed — Subject decision - TP 2 | 11 | 9
Not completed — New therapy for study indication - TP 2 | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | AIN457 6 mg/kg - 3 mg/kg i.v. | Placebo - AIN457 3 mg/kg i.v. | Total
Number analyzed (Participants) | 264 | 262 | 526
Age, Customized [Count of Participants; unit: Participants]
  < 65 years | 253 | 257 | 510
  65 - 75 years | 8 | 4 | 12
  >= 75 years | 3 | 1 | 4
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 99 | 84 | 183
  Male | 165 | 178 | 343
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  White | 180 | 179 | 359
  Black or African American | 7 | 6 | 13
  Asian | 59 | 47 | 106
  American Indian or Alaska Native | 17 | 25 | 42
  Multiple | 1 | 5 | 6
Disease condition [Count of Participants; unit: Participants]
  Ankylosing spondylitis | 208 | 205 | 413
  Non-radiographic axial spondylarthritis | 56 | 57 | 113
Weight [Mean (Standard Deviation); unit: kg] | 77.61 (18.006) | 78.08 (18.444) | 77.85 (18.210)

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants Who Achieved an ASAS40 (Assessment of SpondyloArthritis International Society Criteria)
Description: ASAS40 is ≥ 40% and an absolute improvement from baseline of ≥20 units (range 0-100) in ≥ 3 of the following 4 domains: back pain [10 cm visual analogue scale (VAS)], patient global assessment of disease activity (10 cm VAS), physical function (BASFI; range 0-100) and inflammation (mean score of items 5 and 6 of the BASDAI; both 10 cm VAS) without any worsening in the remaining domain.
  ASAS consists of 6 domains (4 main and 2 additional): 1. Patient's global assessment measured on a visual analog scale (VAS); 2. Patient's assessment of back pain, measured on a VAS; 3. Function represented by Bath Ankylosing Spondylitis Functional Index (BASFI) measured by VAS; 4. Inflammation represented by mean duration and severity of morning stiffness, on the BAS Disease Activity Index (BASDAI) as measured by VAS; 5. Spinal mobility represented by the BAS Metrology Index (BASMI) lateral spinal flexion assessment; 6. C-reactive protein (acute phase reactant).
Time Frame: Baseline to Week 16
Population: Full analysis set with missing responses for any reason imputed as non-responders.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | AIN457 6 mg/kg - 3 mg/kg i.v. | Placebo - AIN457 3 mg/kg i.v.
Number analyzed (Participants) | 264 | 262
percentage of participants | 40.85 [34.94 to 46.76] | 22.94 [17.86 to 28.02]
Statistical Analysis 1: Comparison: AIN457 6 mg/kg - 3 mg/kg i.v. vs Placebo - AIN457 3 mg/kg i.v; Week 16; Test type: Superiority; p < 0.0001, Regression, Logistic; Marginal difference = 17.91, 95% CI 2-sided [10.12 to 25.71]

2. Secondary Outcome: Percentage of Participants Who Achieved Ankylosing Spondylitis Disease Activity Score (ASDAS)-C-Reactive Protein (CRP) Major Improvement
Description: ASDAS-CRP was utilized to assess disease activity status. Parameters used for the ASDAS included: total back pain (BASDAI question 2), patient's global assessment of disease activity, peripheral pain/swelling (BASDAI question 3), duration of morning stiffness (BASDAI question 6) and CRP in mg/L. Disease activity states: inactive disease, moderate disease activity, high disease activity, and very high disease activity. The three values selected to separate these states are: < 1.3 between inactive disease and moderate disease activity; < 2.1 between moderate disease activity and high disease activity; and > 3.5 between high disease activity and very high disease activity. Selected cutoffs for improvement scores are a change of ≥ 1.1 unit for "minimal clinically important improvement" and a change of ≥ 2.0 units for "major improvement" .
Time Frame: Baseline to Week 16
Population: Full analysis set with missing responses for any reason imputed as non-responders.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | AIN457 6 mg/kg - 3 mg/kg i.v. | Placebo - AIN457 3 mg/kg i.v.
Number analyzed (Participants) | 264 | 262
percentage of participants | 27.99 [22.86 to 33.12] | 7.54 [4.44 to 10.64]
Statistical Analysis 1: Comparison: AIN457 6 mg/kg - 3 mg/kg i.v. vs Placebo - AIN457 3 mg/kg i.v; Test type: Superiority; p < 0.0001, Regression, Logistic; Marginal difference = 20.45, 95% CI 2-sided [14.45 to 26.44]

3. Secondary Outcome: The Change From Baseline in Total Bath Ankylosing Spondylitis Disease Activity Index (BASDAI)
Description: BASDAI consists of a 0 through 10 scale (0 indicating no problem and 10 indicating the worst problem, captured as a continuous VAS), which was used to answer six questions pertaining to the five major symptoms of AS: fatigue, spinal pain, peripheral joint pain / swelling,, areas of localized tenderness (enthesitis, or inflammation of tendons and ligaments), morning stiffness duration, morning stiffness severity.
  To give each symptom equal weight, the mean of the two scores relating to morning stiffness is taken into account (questions 5 and 6). The resulting 0 to 10 score is added to the scores for questions 1 through 4. The resulting 0 to 50 score is divided by 5 to give a final 0 10 BASDAI score.
Time Frame: Baseline to Week 16
Population: Full analysis set
Measure: Least Squares Mean (Standard Error); unit: scores on a scale
Arm/Group | AIN457 6 mg/kg - 3 mg/kg i.v. | Placebo - AIN457 3 mg/kg i.v.
Number analyzed (Participants) | 253 | 247
scores on a scale | -2.70 (0.144) | -1.69 (0.144)
Statistical Analysis 1: Comparison: AIN457 6 mg/kg - 3 mg/kg i.v. vs Placebo - AIN457 3 mg/kg i.v; Week 16; Test type: Superiority; p < 0.0001, Mixed Models Analysis; LS mean change = -1.01, 95% CI 2-sided [-1.38 to -0.64], Standard Error of Mean 0.189

4. Secondary Outcome: Percentage of Participants Who Achieved an ASAS 5/6 (Assessment of Spondylarthritis International Society Criteria)
Description: The ASAS 5/6 improvement criteria is an improvement of ≥20% in at least five of all six domains. A higher score on the VAS signifies higher severity.
  ASAS consists of 6 domains (4 main and 2 additional): 1. Patient's global assessment measured on a visual analog scale (VAS); 2. Patient's assessment of back pain, measured on a VAS; 3. Function represented by Bath Ankylosing Spondylitis Functional Index (BASFI) measured by VAS; 4. Inflammation represented by mean duration and severity of morning stiffness, on the BAS Disease Activity Index (BASDAI) as measured by VAS; 5. Spinal mobility represented by the BAS Metrology Index (BASMI) lateral spinal flexion assessment; 6. C-reactive protein (acute phase reactant).
Time Frame: Baseline to Week 16
Population: Full analysis set with missing responses for any reason imputed as non-responders.
Measure: Number (95% Confidence Interval); unit: Percentage of participaants
Arm/Group | AIN457 6 mg/kg - 3 mg/kg i.v. | Placebo - AIN457 3 mg/kg i.v.
Number analyzed (Participants) | 264 | 262
Percentage of participaants | 43.92 [37.94 to 49.90] | 21.77 [16.77 to 26.77]
Statistical Analysis 1: Comparison: AIN457 6 mg/kg - 3 mg/kg i.v. vs Placebo - AIN457 3 mg/kg i.v; Test type: Superiority; p < 0.0001, Regression, Logistic; Marginal difference = 22.15, 95% CI 2-sided [14.36 to 29.95]

5. Secondary Outcome: The Change From Baseline in Total Bath Ankylosing Spondylitis Functional Index (BASFI)
Description: The BASFI is a set of 10 questions designed to determine the degree of functional limitation in subjects with AS. The questions were chosen on the basis of predominant input from subjects with AS. The first eight questions consider activities related to functional anatomy. The final two questions assess the subjects' ability to cope with everyday life. A 0-10 scale (captured as a continuous VAS) is used to answer the questions. The BASFI score is the mean of the ten scales - a value between 0 and 10.
Time Frame: Baseline to Week 16
Population: Full analysis set
Measure: Least Squares Mean (Standard Error); unit: scores on a scale
Arm/Group | AIN457 6 mg/kg - 3 mg/kg i.v. | Placebo - AIN457 3 mg/kg i.v.
Number analyzed (Participants) | 253 | 247
scores on a scale | -2.33 (0.147) | -1.39 (0.148)
Statistical Analysis 1: Comparison: AIN457 6 mg/kg - 3 mg/kg i.v. vs Placebo - AIN457 3 mg/kg i.v; Week 16; Test type: Superiority; p < 0.0001, Mixed Models Analysis; LS mean change = -0.94, 95% CI 2-sided [-1.33 to -0.56], Standard Error of Mean 0.194

6. Secondary Outcome: The Change From Baseline in Short Form-36 Physical Component Summary (SF-36 PCS)
Description: The Short Form-36 Physical Component Summary (SF-36 PCS) is an instrument to measure health-related quality of life among healthy patients and patients with acute and chronic conditions.
  It consists of eight subscales (domains) that can be scored individually: Physical Functioning, Role-Physical, Bodily Pain, General Health, Vitality, Social Functioning, Role- Emotional, and Mental Health. Two overall summary scores, the Physical Component Summary (PCS) and the Mental Component Summary (MCS) also can be computed. The eight domains are based on a scale from 0-100 while PCS and MCS are norm-based scores with a mean of 50 and a standard deviation of 10.
  Higher scores indicate a higher level of functioning. A positive change from baseline score indicates an improvement.
Time Frame: Baseline to Week 16
Population: Full analysis set
Measure: Least Squares Mean (Standard Error); unit: scores on a scale
Arm/Group | AIN457 6 mg/kg - 3 mg/kg i.v. | Placebo - AIN457 3 mg/kg i.v.
Number analyzed (Participants) | 254 | 247
scores on a scale | 7.70 (0.473) | 4.69 (0.473)
Statistical Analysis 1: Comparison: AIN457 6 mg/kg - 3 mg/kg i.v. vs Placebo - AIN457 3 mg/kg i.v; Week 16; Test type: Superiority; p < 0.0001, Mixed Models Analysis; LS mean change = 3.01, 95% CI 2-sided [1.80 to 4.22], Standard Error of Mean 0.615

7. Secondary Outcome: The Change From Baseline in Ankylosing Spondylitis Quality of Life (ASQol)
Description: The ASQoL is a self-administered questionnaire designed to assess health-related quality of life in adult subjects with AS. The ASQoL contains 18 items with a dichotomous yes/no response option. A single point is assigned for each "yes" response and no points for each "no" response, resulting in overall scores that range from 0 (least severity) to 18 (highest severity). As such, lower scores indicate better quality of life. Items include an assessment of mobility/energy, self care and mood/emotion. The recall period is "at the moment".
Time Frame: Baseline to Week 16
Population: Full analysis set
Measure: Least Squares Mean (Standard Error); unit: scores on a scale
Arm/Group | AIN457 6 mg/kg - 3 mg/kg i.v. | Placebo - AIN457 3 mg/kg i.v.
Number analyzed (Participants) | 254 | 247
scores on a scale | -4.65 (0.291) | -2.88 (0.290)
Statistical Analysis 1: Comparison: AIN457 6 mg/kg - 3 mg/kg i.v. vs Placebo - AIN457 3 mg/kg i.v; Week 16; Test type: Superiority; p < 0.0001, Mixed Models Analysis; LS mean change = -1.77, 95% CI 2-sided [-2.51 to -1.04], Standard Error of Mean 0.373

8. Secondary Outcome: The Change From Baseline in High Sensitivity C-Reactive Protein (hsCRP)
Description: This assessment (laboratory assessment) was performed in order to identify the presence of inflammation, to determine its severity and to monitor the response to treatment. Exponentially transformed LSM, the geometric mean ratio of post-baseline/baseline. A value <1 indicates a reduced CRP
Time Frame: Baseline to Week 16
Population: Full analysis set
Measure: Least Squares Mean (Standard Error); unit: ratio
Arm/Group | AIN457 6 mg/kg - 3 mg/kg i.v. | Placebo - AIN457 3 mg/kg i.v.
Number analyzed (Participants) | 246 | 248
ratio | 0.39 (1.063) | 0.89 (1.062)
Statistical Analysis 1: Comparison: AIN457 6 mg/kg - 3 mg/kg i.v. vs Placebo - AIN457 3 mg/kg i.v; Week 16; Test type: Superiority; p < 0.0001, Mixed Models Analysis; Relative LS mean change = 0.44, 95% CI 2-sided [0.37 to 0.51]

9. Secondary Outcome: Percentage of Participants Who Achieved an ASAS20 (Assessment of SpondyloArthritis International Society Criteria)
Description: The ASAS Response Criteria (ASAS20) is defined as an improvement of ≥20% and ≥1 unit on a scale of 10 in at least three of the four main domains and no worsening of ≥20% and ≥1 unit on a scale of 10 in the remaining domain. A higher score on the VAS signifies higher severity.
  ASAS consists of 6 domains (4 main and 2 additional): 1. Patient's global assessment measured on a visual analog scale (VAS); 2. Patient's assessment of back pain, measured on a VAS; 3. Function represented by Bath Ankylosing Spondylitis Functional Index (BASFI) measured by VAS; 4. Inflammation represented by mean duration and severity of morning stiffness, on the BAS Disease Activity Index (BASDAI) as measured by VAS; 5. Spinal mobility represented by the BAS Metrology Index (BASMI) lateral spinal flexion assessment; 6. C-reactive protein (acute phase reactant).
Time Frame: Baseline to Week 16
Population: Full analysis set with missing responses for any reason imputed as non-responders.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | AIN457 6 mg/kg - 3 mg/kg i.v. | Placebo - AIN457 3 mg/kg i.v.
Number analyzed (Participants) | 264 | 262
percentage of participants | 63.94 [58.19 to 69.70] | 40.53 [34.62 to 46.44]
Statistical Analysis 1: Comparison: AIN457 6 mg/kg - 3 mg/kg i.v. vs Placebo - AIN457 3 mg/kg i.v; Test type: Superiority; p < 0.0001, Regression, Logistic; Marginal difference = 23.41, 95% CI 2-sided [15.61 to 31.66]

10. Secondary Outcome: The Percentage of Participants Achieving Ankylosing Spondylitis Disease Activity Score (ASDAS)-C-Reactive Protein (CRP) Inactive Disease.
Description: ASDAS-CRP was utilized to assess disease activity status. Parameters used for the ASDAS included: total back pain (BASDAI question 2), patient's global assessment of disease activity, peripheral pain/swelling (BASDAI question 3), duration of morning stiffness (BASDAI question 6) and CRP in mg/L.
  Disease activity states: inactive disease, moderate disease activity, high disease activity, and very high disease activity. The three values selected to separate these states are: < 1.3 between inactive disease and moderate disease activity; < 2.1 between moderate disease activity and high disease activity; and > 3.5 between high disease activity and very high disease activity. Selected cutoffs for improvement scores are a change of ≥ 1.1 unit for "minimal clinically important improvement" and a change of ≥ 2.0 units for "major improvement"
Time Frame: Baseline to Week 16
Population: Full analysis set with missing responses for any reason imputed as non-responders.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | AIN457 6 mg/kg - 3 mg/kg i.v. | Placebo - AIN457 3 mg/kg i.v.
Number analyzed (Participants) | 264 | 262
percentage of participants | 15.66 [11.53 to 19.78] | 3.08 [1.00 to 5.15]
Statistical Analysis 1: Comparison: AIN457 6 mg/kg - 3 mg/kg i.v. vs Placebo - AIN457 3 mg/kg i.v; Week 16; Test type: Superiority; p < 0.0001, Regression, Logistic; Marginal difference = 12.58, 95% CI 2-sided [7.96 to 17.19]

11. Secondary Outcome: Percentage of Participants Who Achieved ASAS20 (Assessment of Spondylarthritis International Society Criteria) Partial Remission.
Description: ASAS partial remission criteria are defined as a value not above 2 units in each of the four main ASAS domains on a scale of 0-10.
  ASAS consists of 6 domains (4 main and 2 additional): 1. Patient's global assessment measured on a visual analog scale (VAS); 2. Patient's assessment of back pain, measured on a VAS; 3. Function represented by Bath Ankylosing Spondylitis Functional Index (BASFI) measured by VAS; 4. Inflammation represented by mean duration and severity of morning stiffness, on the BAS Disease Activity Index (BASDAI) as measured by VAS; 5. Spinal mobility represented by the BAS Metrology Index (BASMI) lateral spinal flexion assessment; 6. C-reactive protein (acute phase reactant).
Time Frame: Baseline to Week 16
Population: Full analysis set with missing responses for any reason imputed as non-responders.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | AIN457 6 mg/kg - 3 mg/kg i.v. | Placebo - AIN457 3 mg/kg i.v.
Number analyzed (Participants) | 264 | 262
percentage of participants | 14.76 [10.49 to 19.03] | 4.20 [1.77 to 6.63]
Statistical Analysis 1: Comparison: AIN457 6 mg/kg - 3 mg/kg i.v. vs Placebo - AIN457 3 mg/kg i.v; Test type: Superiority; p < 0.0001, Regression, Logistic; Marginal difference = 10.56, 95% CI 2-sided [5.64 to 15.47]

12. Secondary Outcome: Change From Baseline in Pittsburgh Sleep Quality Index (PSQI)
Description: The PSQI is a self-report questionnaire that assesses sleep quality over a 1-month time interval. Consisting of 19 items, the PSQI measures several different aspects of sleep, offering seven component scores and one composite score. The component scores consist of subjective sleep quality, sleep latency (i.e., how long it takes to fall asleep), sleep duration, habitual sleep efficiency (i.e., the percentage of time in bed that one is asleep), sleep disturbances, use of sleeping medication, and daytime dysfunction.
  Each item is weighted on a 0-3 interval scale. The global PSQI score is then calculated by totaling the seven component scores, providing an overall score ranging from 0 to 21, where lower scores denoted a healthier sleep quality.
Time Frame: Baseline to Week 16
Population: Full analysis set
Measure: Least Squares Mean (Standard Error); unit: scores on a scale
Arm/Group | AIN457 6 mg/kg - 3 mg/kg i.v. | Placebo - AIN457 3 mg/kg i.v.
Number analyzed (Participants) | 249 | 246
scores on a scale | -2.42 (0.222) | -1.76 (0.221)
Statistical Analysis 1: Comparison: AIN457 6 mg/kg - 3 mg/kg i.v. vs Placebo - AIN457 3 mg/kg i.v; Test type: Superiority; p = 0.0234, Regression, Logistic; LS mean change = -0.66, 95% CI 2-sided [-1.24 to -0.09], Standard Error of Mean 0.292

ADVERSE EVENTS:
Time Frame: Adverse events were reported for a maximum of 478 days for participants on AIN457 (including placebo switchers) and 182 days for participants on placebo which includes the 84 days in safety follow up.
Description: Any subjects randomized to Placebo were counted under 'Placebo' before being switched to AIN457 and under 'Any AIN457' after being switched to AIN457. It was pre-specified in the Study Protocol to monitor/assess Adverse Events irrespective of AIN457 dose level.
Groups:
- Any AIN457: Participants received secukinumab (AIN457) 6 mg/kg i.v. at baseline, followed by secukinumab 3 mg/kg i.v. every four weeks starting at Week 4 through Week 48 (exposure through Week 52); placebo participants who switched at Week 16 received secukinumab 3 mg/kg i.v. every four weeks starting at Week 16 through Week 48 (exposure through Week 52)
- Placebo Until Week 16: Participants received i.v. placebo at baseline visit), Weeks 4, 8, and 12 , followed by the administration of secukinumab 3 mg/kg i.v. at Week 16 and every four weeks through Week 48 (exposure through Week 52
Arm/Group | Any AIN457 | Placebo Until Week 16
All-Cause Mortality (participants affected / at risk) | 1/517 | 0/261
Serious Adverse Events (participants affected / at risk) | 32/517 | 3/261
Other Adverse Events (participants affected / at risk) | 172/517 | 35/261
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Any AIN457 (N=517) | Placebo Until Week 16 (N=261)
Anaemia (Blood and lymphatic system disorders) | 1 | 0
Acute left ventricular failure (Cardiac disorders) | 1 | 0
Coronary artery occlusion (Cardiac disorders) | 1 | 0
Myocardial infarction (Cardiac disorders) | 2 | 0
Tachycardia (Cardiac disorders) | 1 | 0
Tympanic membrane perforation (Ear and labyrinth disorders) | 1 | 0
Choroiditis (Eye disorders) | 1 | 0
Abdominal pain (Gastrointestinal disorders) | 2 | 0
Colitis (Gastrointestinal disorders) | 1 | 0
Colitis ulcerative (Gastrointestinal disorders) | 2 | 0
Crohn's disease (Gastrointestinal disorders) | 1 | 0
Small intestinal obstruction (Gastrointestinal disorders) | 1 | 0
Chest pain (General disorders) | 1 | 0
Non-cardiac chest pain (General disorders) | 1 | 0
Cholecystitis (Hepatobiliary disorders) | 0 | 1
Drug hypersensitivity (Immune system disorders) | 1 | 0
Anal abscess (Infections and infestations) | 1 | 0
Appendicitis (Infections and infestations) | 1 | 0
COVID-19 pneumonia (Infections and infestations) | 1 | 0
Cellulitis (Infections and infestations) | 2 | 0
Dengue fever (Infections and infestations) | 1 | 0
Lower respiratory tract infection (Infections and infestations) | 1 | 0
Parainfluenzae virus infection (Infections and infestations) | 1 | 0
Pneumonia (Infections and infestations) | 1 | 0
Sepsis (Infections and infestations) | 1 | 0
Tonsillitis (Infections and infestations) | 0 | 1
Hand fracture (Injury, poisoning and procedural complications) | 1 | 0
Lower limb fracture (Injury, poisoning and procedural complications) | 1 | 0
Stab wound (Injury, poisoning and procedural complications) | 0 | 1
Weight decreased (Investigations) | 1 | 0
Fistula (Musculoskeletal and connective tissue disorders) | 1 | 0
Breast cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Seminoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Depression suicidal (Psychiatric disorders) | 1 | 0
Ovarian cyst ruptured (Reproductive system and breast disorders) | 0 | 1
Asthma (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Dermatitis atopic (Skin and subcutaneous tissue disorders) | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 2% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Any AIN457 (N=517) | Placebo Until Week 16 (N=261)
Diarrhoea (Gastrointestinal disorders) | 18 | 5
Nausea (Gastrointestinal disorders) | 12 | 2
COVID-19 (Infections and infestations) | 65 | 10
Nasopharyngitis (Infections and infestations) | 32 | 7
Pharyngitis (Infections and infestations) | 13 | 1
Rhinitis (Infections and infestations) | 11 | 2
Upper respiratory tract infection (Infections and infestations) | 22 | 6
Urinary tract infection (Infections and infestations) | 11 | 1
Arthralgia (Musculoskeletal and connective tissue disorders) | 20 | 1
Headache (Nervous system disorders) | 17 | 9

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The terms and conditions of Novartis' agreements with its investigators may vary. However, Novartis does not prohibit any investigator from publishing. Any publications from a single-site are postponed until the publication of the pooled data (i.e., data from all sites) in the clinical trial.

DOCUMENTS (2):
  • Study Protocol (2019-08-16): https://cdn.clinicaltrials.gov/large-docs/20/NCT04156620/Prot_000.pdf
  • Statistical Analysis Plan (2023-01-12): https://cdn.clinicaltrials.gov/large-docs/20/NCT04156620/SAP_001.pdf